CLINICAL TRIAL: NCT02751788
Title: Physical Activity and Screen-Time Regulations in Childcare Centers: Influence on Young Children's Health Behaviors (Pause & Play) - Aim 1
Brief Title: Physical Activity and Screen-Time Regulations in Childcare Centers - Aim 1
Acronym: Pause and Play
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Amanda Staiano, PBRC Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2015-044
Record Dates: First submitted 2016-04-19; First posted 2016-04-26 (Estimated); Results first posted 2023-09-07 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Childhood Obesity
Keywords: childcare center regulations; physical activity; sedentary behavior; screen-time behavior
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this project is to examine the physical activity and screen-time environment of licensed childcare centers before and after the enactment of new state regulations.

DETAILED DESCRIPTION:
Pause and Play will take a prospective observational epidemiological approach before and after enactment of new regulations. 10 childcare centers licensed in East Baton Rouge Parish will be randomly selected and standardized behavioral observation scales will be used to objectively quantify the physical activity and screen-time environment of the centers and the children's behaviors both in and outside the center. These assessments will be collected twice during the 2-year grant period to capture potential changes after the policies are implemented.

ELIGIBILITY:
Inclusion Criteria:

* Licensed by DOE as a Class A or Class B childcare center
* Located in East Baton Rouge Parish
* Current childcare enrollment of at least 18 children between the ages of 3-4 years

Exclusion Criteria:

* Childcare center and/or childcare center director unwilling to participate

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Ten licensed DOE Class A or B childcare centers will be randomly selected from a list of all DOE licensed childcare centers in East Baton Rouge Parish (EBR)
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Staiano, PhD, Principal Investigator — PBRC Assistant Professor
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kracht CL, Webster EK, Staiano AE. A natural experiment of state-level physical activity and screen-time policy changes early childhood education (ECE) centers and child physical activity. BMC Public Health. 2020 Mar 24;20(1):387. doi: 10.1186/s12889-020-08533-8. PMID 32209069
- [Result] Staiano AE, Webster EK, Allen AT, Jarrell AR, Martin CK. Screen-Time Policies and Practices in Early Care and Education Centers in Relationship to Child Physical Activity. Child Obes. 2018 Aug/Sep;14(6):341-348. doi: 10.1089/chi.2018.0078. PMID 30199286
- [Result] Staiano AE, Allen AT, Fowler W, Gustat J, Kepper MM, Lewis L, Martin CK, Romain JS, Webster EK. State Licensing Regulations on Screen Time in Childcare Centers: An Impetus for Participatory Action Research. Prog Community Health Partnersh. 2018;12(1S):101-109. doi: 10.1353/cpr.2018.0025. PMID 29755053
- [Result] Joseph ED, Kracht CL, St Romain J, Allen AT, Barbaree C, Martin CK, Staiano AE. Young Children's Screen Time and Physical Activity: Perspectives of Parents and Early Care and Education Center Providers. Glob Pediatr Health. 2019 Jul 24;6:2333794X19865856. doi: 10.1177/2333794X19865856. eCollection 2019. PMID 31384633
- [Result] Webster EK, Martin CK, Staiano AE. Fundamental motor skills, screen-time, and physical activity in preschoolers. J Sport Health Sci. 2019 Mar;8(2):114-121. doi: 10.1016/j.jshs.2018.11.006. Epub 2018 Nov 24. PMID 30997257
- [Result] Martins, C., Webster, E. K., Bandeira, P. F. R., & Staiano, A. E. (2022). Identifying Fundamental Motor Skills Building Blocks in Preschool Children From Brazil and the United States: A Network Analysis. Journal of Motor Learning and Development, 10(1), 96-115. Retrieved Mar 27, 2024, from https://doi.org/10.1123/jmld.2021-0022
- [Result] Kracht CL, Webster EK, Staiano AE. Relationship between the 24-Hour Movement Guidelines and fundamental motor skills in preschoolers. J Sci Med Sport. 2020 Dec;23(12):1185-1190. doi: 10.1016/j.jsams.2020.06.021. Epub 2020 Jul 5. PMID 32653249
- [Result] Kracht CL, Webster EK, Staiano AE. Sociodemographic Differences in Young Children Meeting 24-Hour Movement Guidelines. J Phys Act Health. 2019 Oct 1;16(10):908-915. doi: 10.1123/jpah.2019-0018. Epub 2019 Sep 6. PMID 31491748

RESULTS

PARTICIPANT FLOW:
Groups:
- ECE Center Changes and Changes in Child Physical Activity: Aim 1 of this study was to evaluate the association among ECE center changes in practices, environment, staff behaviors, and policies, and changes in child physical activity and sedentary behavior while attending the ECE centers.
Period: Overall Study
Arm/Group | ECE Center Changes and Changes in Child Physical Activity
Started | 112
Completed | 49
Not Completed | 63

BASELINE CHARACTERISTICS:
Arm/Group | ECE Center Changes and Changes in Child Physical Activity
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 37
  Race: African American | 7
  Race: Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Environment and Policy Assessment and Observation (EPAO) Score and EPAO Subscales.
Description: The EPAO instrument will be used, which is a comprehensive, day-long observation that objectively defines the nutrition and physical activity environmental characteristics of child care centers. To address the specific aim, only the EPAO variables related to physical activity and screen-time will be included in the assessment. Means, standard deviations, and Pearson correlations will be calculated to describe the sample and examine relationships among the environment subscales at baseline and follow-up. Differences in center characteristics (i.e. racial distribution) will be tested using t-tests and chi-square tests. Repeated measures analysis of covariance (ANCOVAs) will be used to examine change in the EPAO score overall. Higher scores indicate higher compliance with best practices.
Time Frame: 1 year
Measure: Mean (Standard Error); unit: minutes
Arm/Group | ECE Center Changes and Changes in Child Physical Activity
Number analyzed (Participants) | 112
minutes
  Active Play (minutes) | -.12 (.05)
  Television viewing (minutes) | .21 (.28)
  Non-television screen-time (minutes) | .25 (.10)
  Television screen-time (minutes) | .21 (.11)

2. Secondary Outcome: Changes in Practice-based Survey Items Based on Childcare Director Responses.
Description: A survey will be administered to the director of each childcare center to determine the following: awareness of the new policy; structured programs and/or field trips that allow children to be physically active (including number of times per day or week); if one or more community organizations support or provide physical activity programs at the center; whether or not the childcare center has policies regarding television viewing and computer use; amount of time allowed for free play; and amount of time spent outside.
Time Frame: 1 Year
Population: Ten centers were enrolled in this Study. One site dropped out. The analysis provided is only year two.
Measure: Count of Participants; unit: Participants
Arm/Group | ECE Center Changes and Changes in Child Physical Activity
Number analyzed (Participants) | 10
Participants
  Awareness of new policy (Year 2): number analyzed (Participants) | 9
  Awareness of new policy (Year 2): Yes | 7
  Awareness of new policy (Year 2): No | 2
  Field Trips (Year 2): number analyzed (Participants) | 9
  Field Trips (Year 2): Yes | 5
  Field Trips (Year 2): No | 4
  Community organizations - provide physical activity programs (Year 2): number analyzed (Participants) | 9
  Community organizations - provide physical activity programs (Year 2): Yes | 3
  Community organizations - provide physical activity programs (Year 2): No | 6
  Children are not allowed any screen time at the center (Year 2): number analyzed (Participants) | 9
  Children are not allowed any screen time at the center (Year 2): Yes | 4
  Children are not allowed any screen time at the center (Year 2): No | 5
  Children are allowed at least 60 minutes of free play (Year 2): number analyzed (Participants) | 9
  Children are allowed at least 60 minutes of free play (Year 2): Yes | 9
  Children are allowed at least 60 minutes of free play (Year 2): No | 0
  Children are allowed at least 90 minutes of outdoor time (Year 2): number analyzed (Participants) | 9
  Children are allowed at least 90 minutes of outdoor time (Year 2): Yes | 5
  Children are allowed at least 90 minutes of outdoor time (Year 2): No | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | ECE Center Changes and Changes in Child Physical Activity
All-Cause Mortality (participants affected / at risk) | 0/112
Serious Adverse Events (participants affected / at risk) | 0/112
Other Adverse Events (participants affected / at risk) | 0/112

LIMITATIONS AND CAVEATS:
The timing of some assessments occurred into 2017 due to delays, there's a chance ECE centers changed their policy after the regulations were first released thus the baseline data collection was not a true baseline. However, this study did utilize handbooks for policy scoring & baseline policies were dated for the 2016-2017 school year. Another limitation is that ECE centers were aware of the day of observation, there's a potential the center made changes to present as a healthier environment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT02751788/Prot_SAP_000.pdf